CLINICAL TRIAL: NCT01711372
Title: Predictive Executive Functioning Models Using Interactive Tangible-Graphical Interface Devices, Phase 2 Trials
Brief Title: Predictive Executive Functioning Models Using Interactive Tangible-Graphical Interface Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CogCubed, Corp (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 131209-12
Record Dates: First submitted 2012-10-16; First posted 2012-10-22 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Patients were those with ADHD and age and gender matched controls who completed a game placed on Sifteo cubes to assess for ADHD. The intervention was a game to screen for ADHD.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The person having the patient play the came did not know if the patient had ADHD or not.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controls who played Groundskeeper game (Placebo Comparator): Controls played a go/no go task on Sifteo cubes to asses for attentional capabilities.
  Interventions: Device: Groundskeeper game for controls
- Probands played groundskeeper game (Active Comparator): Patients with ADHD played a go/no go task on Sifteo cubes to asses for attentional capabilities
  Interventions: Device: Groundskeeper game for ADHD

INTERVENTIONS:
Device: Groundskeeper game for controls — The Groundskeeper game is a go/no go task that captures reaction time and movement using the accelerometers and touch capabilities of the Sifteo cubes.
  Arms: Controls who played Groundskeeper game
Device: Groundskeeper game for ADHD — The Groundskeeper game is a go/no go task that captures reaction time and movement using the accelerometers and touch capabilities of the Sifteo cubes.
  Arms: Probands played groundskeeper game

SUMMARY:
A new company called CogCubed has created a new game based on the Sifteo Cube (http://www.sifteo.com) platform. These new hands-on digitized cubes are unique, motion-sensitive wireless blocks that contain multiple sensors that can interact with one another. CogCubed is providing the data for this study. The game will be played in a 30 minute sessions by subjects ages 6-17. Subjects recruited to play the game will be those with ADHD and those without, matched by gender and age. Those with comorbidities of developmental delay, mental retardation, psychosis, schizophrenia, bipolar disorder and substance use disorders will be excluded, as well as any physiological disability that affects upper limb movement and/or coordination. Informed consent will be obtained from parents and patient prior to administering the game. Parents will fill out a Conner's Brief Rating Scale and a Conner's Brief Rating Scale, Teacher's version will also be supplied to be filled out at school. The hypothesis is that by analyzing data generated from this new gaming platform named Sifteo for which a game was created, which uses auditory and visual stimuli and distracters, the investigators expect that they will be able to provide a more accurate profile of impulsivity and inattention.

DETAILED DESCRIPTION:
Current diagnostic aids used in treating ADHD are currently expensive, time intensive, and provide little information about accessory movements in response to a stimulus. One in ten children, ages 5 to 17, has been diagnosed with ADHD.

Tests such as the Conners' Rating Scale require subjective responses from parents and teachers, making coordination difficult. The computerized Conners' Continuous Performance Test (CPT) provides objective data in regards to inattention and impulsive patterns of response. However, it does not provide data regarding accessory movements such as restlessness, hyperactivity, and other inappropriate movements. If the subject taking the exam has a reading disorder, it will impair his or her ability to respond accurately and it will increase response time. The T.O.V.A. is another computer based test used as a diagnostic aid for ADHD, which uses a microswitch to record responses. It does utilize auditory and visual stimuli, which removes the reading level limitation. However, it is unable to measure to measure accessory movements that may be contributing to reaction time and errors of omission and commission.

Because of these limitations, a new company called CogCubed has created a new game based on the Sifteo Cube (http://www.sifteo.com) platform. These new hands-on digitized cubes are unique, motion-sensitive wireless blocks that contain multiple sensors that can interact with one another. CogCubed is providing the data for this study. The game will be played in a 30 minute sessions by subjects ages 6-17. Subjects recruited to play the game will be those with ADHD and those without, matched by gender and age. Those with comorbidities of developmental delay, mental retardation, psychosis, schizophrenia, bipolar disorder and substance use disorders will be excluded, as well as any physiological disability that affects upper limb movement and/or coordination. Informed consent will be obtained from parents and patient prior to administering the game. Parents will fill out a Conner's Brief Rating Scale and a Conner's Brief Rating Scale, Teacher's version will also be supplied to be filled out at school.

The hypothesis is that by analyzing data generated from this new gaming platform named Sifteo for which a game was created, which uses auditory and visual stimuli and distracters, the investigators expect that they will be able to provide a more accurate profile of impulsivity and inattention. The investigators expect that inattention will have more errors of omission and less tilt movements than control and impulsivity will be represented as more commission and greater tilting movements than control. This trial builds on the previous results of our phase 1 trials used to create the predictive algorithms to analyze the data and predict the likelihood of ADHD diagnosis based on patterns of game play behavior.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17, males and females
* Individuals with ADHD
* Individuals without ADHD
* Depressive Disorders
* Anxiety Disorders
* Oppositional Defiant Disorder
* Panic Disorder
* Eating Disorder

Exclusion Criteria:

* Developmental Delay
* IQ below 70
* Low functioning Autism Spectrum Disorders
* Psychosis
* Substance Use Disorders
* Medical comorbidities that involve any motoric disability that affects upper-limb movement and/or strength

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2016-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika D Roots, MD, Principal Investigator — CogCubed, Corp; Jaideep Srivastava, PhD, Principal Investigator — CogCubed, Corp
Locations (2):
- United States (2):
  - Groves Academy, Saint Louis Park, Minnesota
  - Egli Assessment, Waconia, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Faraone SV, Newcorn JH, Antshel KM, Adler L, Roots K, Heller M. The Groundskeeper Gaming Platform as a Diagnostic Tool for Attention-Deficit/Hyperactivity Disorder: Sensitivity, Specificity, and Relation to Other Measures. J Child Adolesc Psychopharmacol. 2016 Oct;26(8):672-685. doi: 10.1089/cap.2015.0174. Epub 2016 Apr 22. PMID 27105181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Invited for participation consecutive patients referred to a child psychiatrist. From this cohort of patients, two groups formed. Patients who had received ADHD diagnosed and those who had not.
Pre-assignment Details: 113 patients were screened for ADHD vs no ADHD. Those with ADHD were asked to not take stimulant medications for at least 3 days prior to participating. Company no longer exists and no longer has access to data collected. Only information in published study results available.
Groups:
- ADHD Group: Patients with ADHD played a go/no go task on Sifteo cubes to assess for attentional capabilities. Groundskeeper Game: The Groundskeeper game is a go/no-go task that captures reaction time and movement using the accelerometers and touch capabilities on the Sanvello cubes.
- Control Group: Controls played a go/no go task on Sifteo cubes to assess for attentional capabilities. Groundskeeper Game: The Groundskeeper game is a go/no-go task that captures reaction time and movement using the accelerometers and touch capabilities on the Sanvello cubes.
Period: Overall Study
Arm/Group | ADHD Group | Control Group
Started | 66 | 47
Completed | 66 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The patients who completed all screening tests and intervention for this trial were 113 patients. Company no longer exists. Only information in published study results available.
Groups:
- ADHD Group: Patients with ADHD played a go/no go task on Sifteo cubes to asses for attentional capabilities.
  Groundskeeper Game: The Groundskeeper game is a go/no go task that captures reaction time and movement using the accelerometers and touch capabilities of the Sifteo cubes.
- Control Group: Controls played a go/no go task on Sifteo Cubes to asses for attentional capabilities.
  Groundskeeper Game: The Groundskeeper game is a go/no go task that captures reaction time and movement using the accelerometers and touch capabilities of the Sifteo cubes.
- Total: Total of all reporting groups
Arm/Group | ADHD Group | Control Group | Total
Number analyzed (Participants) | 66 | 47 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 66 | 47 | 113
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 38 | 18 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 58 | 38 | 96
  Other | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 66 | 47 | 113
Psychiatric Disorders [Count of Participants; unit: Participants]
  Anxiety Disorders | 33 | 45 | 78
  Mood Disorders | 27 | 36 | 63
  Disruptive Behavior Disorders | 11 | 8 | 19
  Autism Spectrum Disorders | 6 | 2 | 8
  Reading Disability | 23 | 10 | 33

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Receiver Operating Characteristic (ROC) Curve- Groundskeeper Game
Description: ROC charts the false-positive (horizontal axis) and the sensitivity or true-positive rate (vertical axis) of the Groundskeeper game at discriminating child psychiatric patients with and without ADHD. Determines diagnostic accuracy of Groundskeeper game for ADHD. For each participant, predicted values were computed from the logistic regression models (correcting for age, sex and medication status). For each successive point on the logit scale sensitivity and specificity of the logit was computed as a predictor of ADHD diagnosis, by predicting those higher than the cut-point to have ADHD and the others not to have ADHD. These data were used to draw the ROC curve. ROC analysis summarized diagnostic efficiency with the area under the curve (AUC) statistic. The AUC ranges from 0.5 (for a diagnostically useless test) to 1.0 (for a diagnostic test that is a perfect predictor).
Time Frame: 30 minutes
Population: Data from both participants with and without ADHD used in calculation of AUC of ROC. Diagnostic accuracy applies to both arm/groups of participants. Company no longer exists. Only information in published study results available.
Measure: Number; unit: Proportion of accurate ADHD Diagnoses
Groups:
- All Participants in the Study With and Without ADHD: Data from both participants with and without ADHD used in calculation of AUC of ROC. Diagnostic accuracy applies to both arm/groups of participants. Company no longer exists. Only information in published study results available.
Arm/Group | All Participants in the Study With and Without ADHD
Number analyzed (Participants) | 113
Proportion of accurate ADHD Diagnoses | 0.78
Statistical Analysis 1: Comparison: All Participants in the Study With and Without ADHD; AUC or ROC for Groundskeeper Game; Test type: Other; Chi-squared; AUC of ROC is 0.78

2. Secondary Outcome: Area Under the Receiver Operating Characteristic (ROC) Curve- Conners Brief Rating Scale Parent Version (Inattention Subscale)
Description: Parent completed the Connors Brief rating Scale Parent Version, with the Inattention subscale extracted for analysis. Scores for this assessment are converted to percentile scores for each age group with higher scores indicating more likelihood of ADHD. ROC charts the false-positive rate (horizontal axis) and the sensitivity or true-positive rate (vertical axis) of discriminating child psychiatric patients with and without ADHD. Determines diagnostic accuracy of Conners Scale for ADHD. ROC analysis summarizes diagnostic efficiency with the area under the curve (AUC) statistic. The AUC ranges from 0.5 (for a diagnostically useless test) to 1.0 (for a diagnostic test that is a perfect predictor).
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Number; unit: Proportion of accurate ADHD Diagnoses
Arm/Group | All Participants in the Study With and Without ADHD
Number analyzed (Participants) | 113
Proportion of accurate ADHD Diagnoses | 0.76
Statistical Analysis 1: Comparison: All Participants in the Study With and Without ADHD; Test type: Other; AUC of ROC. Proportion of accurate ADHD diagnoses is 0.76

3. Secondary Outcome: Area Under the Receiver Operating Characteristic (ROC) Curve- Continuous Performance Task (CPT)
Description: CPT measures sustained attention. Participants were asked to press the space bar whenever any letter except the letter "X: appeared on the computer screen. Used the percent certainty that the CPT II results were in the clinical range in this analysis. ROC charts the false-positive rate (horizontal axis) and the sensitivity or true-positive rate (vertical axis) of discriminating child psychiatric patients with and without ADHD. Determines diagnostic accuracy of Conners scales for ADHD. ROC analysis summarizes diagnostic efficiency with the Area Under the Curve (AUC) statistic. The AUC ranges from 0.5 (for a diagnostically useless test) to 1.0 (for a diagnostic test that is a perfect predictor).
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Number; unit: Proportion of accurate ADHD Diagnoses
Arm/Group | All Participants in the Study With and Without ADHD
Number analyzed (Participants) | 113
Proportion of accurate ADHD Diagnoses | 0.62
Statistical Analysis 1: Comparison: All Participants in the Study With and Without ADHD; Test type: Other — AUC of ROC; AUC of ROC. Proportion of accurate ADHD diagnosis is 0.62

ADVERSE EVENTS:
Time Frame: Company no longer exits. Only information in published study results available. No information available on monitoring/frequency of Adverse Events
Description: Company no longer exits. Only information in published study results available. No information available on monitoring/frequency of Adverse Events
Groups:
- ADHD Group; Control Group: Patient with ADHD played a go/no go task on Sifteo cubes to asses for attentional capabilities.
  Groundskeeper Game: The Groundskeeper game is a go/no go task that captures reaction time and movement using the accelerometers and touch capabilities of the Sifteo Cubes.
Arm/Group | ADHD Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes